CLINICAL TRIAL: NCT04543500
Title: Self-regulation of Prefrontal Cortex During Emotional Cognitive Control
Acronym: SPrC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Robin Aupperle, Principal Investigator, Laureate Institute for Brain Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019-012; F31MH122090 (NIH)
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteers; Cognitive Function

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Left Dorsolateral Prefrontal Cortex rtfMRI-nf (Experimental): Real-time functional magnetic resonance imaging neurofeedback (rtfMRI-nf) will target left dorsolateral prefrontal cortex. Participants in this arm will receive active feedback while attempting to modulate their neural activity during an emotional cognitive control task.
  Interventions: Other: Real-time functional magnetic resonance neurofeedback (rtfMRI-nf)
- Sham Left Dorsolateral Prefrontal Cortex rtfMRI-nf (Active Comparator): Real-time functional magnetic resonance imaging neurofeedback (rtfMRI-nf) will target left postcentral gyrus. Participants in this arm will receive sham feedback while attempting to modulate their neural activity during an emotional cognitive control task.
  Interventions: Other: Real-time functional magnetic resonance neurofeedback (rtfMRI-nf)

INTERVENTIONS:
Other: Real-time functional magnetic resonance neurofeedback (rtfMRI-nf) — Real-time functional magnetic resonance imaging neurofeedback (rtfMRI-nf) is a procedure using an MRI scanner that allows participants to observe their own neural activity in the moment. They are taught to self-regulate this activity during a task.

SUMMARY:
Deficits in emotional cognitive control are present in a number of clinical psychiatric populations including depression, anxiety, and PTSD. Deficits in this domain of function limit one's ability to focus attention on goal directed activities while inhibiting reactions to irrelevant emotional stimuli, and this contributes to the symptoms of these disorders and makes individuals less likely to be successful in existing treatments. The left dorsolateral prefrontal cortex (LDLPFC) and its connectivity with other regions (i.e., dorsal anterior cingulate cortex, ventromedial prefrontal cortex, insula, amygdala) is thought to play a central role in facilitating emotional cognitive control. However, past research has primarily utilized correlational approaches that limit conclusions about the directionality of these relationships. Enhancing our understanding of the neural underpinnings of emotional cognitive control could be valuable for informing treatment for populations with deficits in these processes.

The current study utilizes a neuromodulatory approach called real-time functional magnetic resonance imaging neurofeedback (rtfMRI-nf) whereby participants observe their own neural activity in the moment and are taught to self-regulate this activity. Healthy adult participants will be trained to increase neural activity in LDLPFC while involved in mental tasks involving emotional cognitive control processes. The mental tasks will include counting, remembering words, or planning events while viewing negatively-valenced emotional words (e.g., kill, death, threat). This study will use an experimental approach with participants being randomized to either LDLPFC rtfMRI-nf or control rtfMRI-nf where participants receive neural feedback from a region not involved with emotional cognitive control processes. Resting-state fMRI scans and behavioral testing sessions will take place before and after rtfMRI-nf.

The specific aims are to examine the impact of LDLPFC rtfMRI-nf on: (1) LDLPFC activity during emotional cognitive control and (2) LDLPFC functional connectivity with other brain regions during rest. Additionally, this study will examine the neural correlates of emotional cognitive control independent of rtfMRI-nf. Thus, the final specific aim is to (3) Investigate relationships between individual differences in LDLPFC engagement, cognitive control performance, trauma history, and sleep quality. To facilitate the relevance of these findings to clinical populations, trauma exposure and sleep quality will be explored as moderators of neural change across time for those in the rtfMRI-nf group.

To these ends, this study will use rtfMRI-nf to experimentally investigate the relationship between LDLPFC activity and emotional cognitive control as well as investigate these neural mechanisms independent of rtfMRI-nf. This research will improve our understanding of emotional cognitive control and demonstrate whether this is a modifiable target for intervention in populations with deficits in this domain of function.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* sufficient English proficiency to complete procedures
* absence of any DSM-5 psychiatric disorder

Exclusion Criteria:

* meeting criteria for any DSM-5 psychiatric disorder
* current prescription of psychiatric medication
* history of moderate to severe traumatic brain injury
* diagnosis of neurologic disorders
* current alcohol/drug abuse
* MRI contra-indications (e.g., metal in body)
* uncorrected vision/hearing problems

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-04-16 (Actual); Study Completion 2022-04-16 (Actual)

PRIMARY OUTCOMES:
Left dorsolateral prefrontal cortex activity during emotional cognitive control (pre- to post-neurofeedback) | Approximately 2 hours after baseline assessment
  Individual ability to regulate left dorsolateral prefrontal cortex activity during an emotional cognitive control task will be assessed before and after neurofeedback for both active and sham conditions.

SECONDARY OUTCOMES:
Left dorsolateral prefrontal cortex functional connectivity with other brain regions during rest (pre- to post-neurofeedback) | Approximately 2 hours after baseline assessment
  Individual functional connectivity values between left dorsolateral prefrontal cortex and other brain regions during rest will be assessed before and after neurofeedback for both active and sham conditions.

OTHER OUTCOMES:
Emotional Stroop Average Reaction Time | Approximately 1 day after baseline assessment.
  Average reaction time on the emotion condition of the emotional Stroop task.
Color Word Stroop Average Reaction Time | Approximately 1 day after baseline assessment.
  Average reaction time on the inhibition condition of the color word Stroop task.
Flanker Task Average Reaction Time | Approximately 1 day after baseline assessment.
  Average reaction time on the incongruent condition of the Flanker task.
Emotional Stroop Reaction Time Difference | Approximately 1 day after baseline assessment.
  Difference in reaction time for emotional versus neutral conditions of the emotional Stroop task.
Color Word Stroop Reaction Time Difference | Approximately 1 day after baseline assessment.
  Difference in reaction time for inhibition versus reading conditions of the emotional Stroop task.
Flanker task Reaction Time Difference | Approximately 1 day after baseline assessment.
  Difference in reaction time for incongruent versus congruent conditions of the Flanker task.

CONTACTS AND LOCATIONS:
Overall Officials: Robin L Aupperle, Ph.D., Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers. Following future publication of the data collected from the study, information about analyses and limited data and/or code will be available upon individual request from the authors.